CLINICAL TRIAL: NCT05106517
Title: Attending Physician of Shenzhen People's Hospital
Brief Title: Denosumab vs Zoledronic Acid and Osteoporotic Compression Fracture
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shenzhen People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ShenzhenPH spine wang04
Record Dates: First submitted 2021-10-09; First posted 2021-11-03 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-02

CONDITIONS: Denosumab vs Zoledronate
MeSH Terms: interventions — Denosumab; Injections, Subcutaneous; Zoledronic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- denosumab (Experimental): Denosumab 60mg/6 months subcutaneously + placebo intravenous
  Interventions: Drug: Denosumab
- zoledronic acid (Experimental): intravenous zoledronic acid and placebo /6 months subcutaneously
  Interventions: Drug: Zoledronic acid

INTERVENTIONS:
Drug: Denosumab — Denosumab 60mg/6 months subcutaneously + placebo iv
  Other Names: Denosumab 6 month/subcutaneous
  Arms: denosumab
Drug: Zoledronic acid — Iv zoledronic acid and placebo /6 months subcutaneously
  Other Names: Zoledronic acid intravenous once a year
  Arms: zoledronic acid

SUMMARY:
Bone mineral density and function at 1 year after screw fixation with denosumab vs zoledronic acid for osteoporotic vertebral compression fractures: a parallel double-blind randomized controlled clinical trial

DETAILED DESCRIPTION:
Conduct a single-center, double-blind, randomized controlled clinical trial according to clinical Trial Reporting Standards (CONSORT). Bone mineral density and function of osteoporotic vertebral compression fracture (OVCF) were compared 1 year after screw internal fixation with denosumab vs zoledronic acid in Shenzhen People's Hospital from September, 2021 to November, 2022. The study was approved by Shenzhen People's Hospital and informed consent was signed.

ELIGIBILITY:
Inclusion Criteria:

* Must be age between 40 and 90 years old
* X-ray diagnosis of 1-2 vertebral compression fractures
* Dual eneragy X ray test for bone mineral density T value less than -1
* fracture history lasted within 6 weeks
* Must be MRI showed bone marrow edema of injured segment
* Must be lower back pain, local spines tenderness

Exclusion Criteria:

* Must be able to have no posterior vertebral wall fracture
* Must be able to have no patients with intervertebral fissure
* Must be able to have no infection
* Must be able to have no malignancy
* Must be able to have no neurological dysfunction
* Must be able to have no calcium level ≤2.13 mmol/L
* Must be able to have no previous use of anti-osteoporosis drugs
* Must be able to have no inability to perform magnetic resonance imaging
* Must be able to have no prior back surgery
* Must be able to have no other established contraindications for elective surgery

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 122 (Estimated)
Dates: Start 2021-09-08 (Actual); Primary Completion 2023-03-05 (Estimated); Study Completion 2023-03-11 (Estimated)

PRIMARY OUTCOMES:
age | up to 12 months
  participants age
sex | up to 12 months
  participants sex
height | up to 12 months
  participants height cm
BMI | up to 12 months
  participants body mass index
serum osteocalcin | up to 12 months
  osteocalcin in the N terminal molecular fragment
serum Procollagen type 1 n-terminal propeptide P1NP | up to 12 months
  Procollagen type 1 n-terminal propeptide
serum C-terminal cross-linked type 1 collagen terminal peptide CTX | up to 12 months
  C-terminal cross-linked type 1 collagen terminal peptide
Serum total calcium | up to 12 months
  Serum total calcium level
lumber spine bone mineral density | up to 12 months
  Dual energy X ray for lumber spine bone mineral density
hip bone mineral density | up to 12 months
  DEXA for hip bone mineral density
MRI for lumber | up to 12 months
  Bone marrow edema and adjacent intervertebral disc were detected by MRI
pain visual analogue scores (VAS) | up to 12 months
  pain visual analogue scores (VAS) use categories to differentiate pain intensity. There is a wide variability of terms used to describe each category and the rating may be divided into four (0 -3) or six (0 -5) categories. Patients score their pain intensity from absent (0) to severe (3) or from none (0) to very severe (5)

SECONDARY OUTCOMES:
The Roland-Morris Disability Questionnaire | up to 12 month
  The Roland-Morris Disability Questionnaire is a health status measure designed to be completed by patients to assess physical disability due to low back pain.
QUALEFFO-31 | up to 12 month
  Quality of Life Questionnaire of the European Foundation for Osteoporosis (QUALEFFO) was developed in 1997 to evaluate quality of life for patients with osteoporosis. The questionnaire assesses quality of life in the aspect of pain, physical function, social function, general health, and mental health
EuroQol-5D (EQ-5D) | up to 12 month
  EQ-5D descriptive system is a preference-based HRQL measure with one question for each of the five dimensions that include mobility, self-care, usual activities, pain/discomfort, and anxiety/depression.

CONTACTS AND LOCATIONS:
Locations (1):
- ShenzhenPH, Shenzhen, Guangdong, China

IPD SHARING:
Plan to Share IPD: No